CLINICAL TRIAL: NCT04588480
Title: A PHASE 1/2, PLACEBO-CONTROLLED, RANDOMIZED, AND OBSERVER-BLIND STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A SARS-COV-2 RNA VACCINE CANDIDATE AGAINST COVID-19 IN HEALTHY JAPANESE ADULTS
Brief Title: Study to Evaluate the Safety, Tolerability, and Immunogenicity of an RNA Vaccine Candidate Against COVID-19 in Healthy Japanese Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C4591005
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: SARS-CoV-2 Infection; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BNT162b2 (Experimental): BNT162b2 (intramuscular injection)
  Interventions: Biological: BNT162b2
- Placebo (Placebo Comparator): Placebo (intramuscular injection)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BNT162b2 — BNT162b2 (intramuscular injection)
  Arms: BNT162b2
Other: Placebo — Placebo (intramuscular injection)
  Arms: Placebo

SUMMARY:
This is a Phase 1/2, randomized, placebo-controlled, and observer-blind study in healthy Japanese adults.

The study will evaluate the safety, tolerability, and immunogenicity of the SARS-CoV-2 RNA vaccine candidate against COVID-19:

* As 2 doses, separated by 21 days
* At a single dose level
* In adults 20 to 85 years of age

DETAILED DESCRIPTION:
From protocol amendment 3, this study is transitioned from a clinical trial to a postmarketing study (Phase 4) according to the Japanese regulation, because BNT162b2 was approved by the Ministry of Health, Labour and Welfare on 14 February 2021.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male or female participants between the ages of 20 and 85 years, inclusive, at randomization.
* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for inclusion in the study.
* Capable of giving personal signed informed consent.

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Known infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
* Receipt of medications intended to prevent COVID-19.
* Previous confirmed diagnosis of COVID-19.
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Previous vaccination with any coronavirus vaccine.
* Individuals who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
* Receipt of blood/plasma products or immunoglobulin, from 60 days before study intervention administration or planned receipt throughout the study.
* Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
* Previous participation in other studies involving study intervention containing lipid nanoparticles.
* Subset only: Any screening hematology and/or blood chemistry laboratory value that meets the definition of a ≥ Grade 1 abnormality.
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Japan (2):
  - SOUSEIKAI Sumida Hospital, Sumida-ku, Tokyo
  - SOUSEIKAI PS Clinic, Fukuoka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haranaka M, Baber J, Ogama Y, Yamaji M, Aizawa M, Kogawara O, Scully I, Lagkadinou E, Tureci Ӧ, Sahin U, Dormitzer PR, Gruber WC, Lockhart S. A randomized study to evaluate safety and immunogenicity of the BNT162b2 COVID-19 vaccine in healthy Japanese adults. Nat Commun. 2021 Dec 14;12(1):7105. doi: 10.1038/s41467-021-27316-2. PMID 34907170
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591005

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Originally, study was blinded and participants received 2 doses of ribonucleic acid (RNA)-based COVID-19 vaccine (BNT162b2) and placebo. After protocol amendment 3, the study was unblinded and all participants who originally received placebo were offered the opportunity to receive BNT162b2 vaccine before the 6-month follow-up visit.
Groups:
- BNT162b2: Participants received 2 doses of blinded 30 microgram (mcg) BNT162b2 vaccine as an intramuscular injection separated by 21 days. Participants were followed up to 12 months after last dose of vaccination.
- Placebo: Participants received 2 doses of placebo (normal sterile saline solution) as an intramuscular injection separated by 21 days. Participants were followed up to 12 months after last dose of vaccination.
- Placebo Then BNT162b2: Participants who originally received 2 doses of blinded placebo were administered 2 doses of 30 mcg BNT162b2 vaccine as intramuscular injection separated by 21 days after unblinding. Participants were followed for up to 6 months after last dose of vaccination.
Period: Blinded Phase: Up to 6 Months
Arm/Group | BNT162b2 | Placebo | Placebo Then BNT162b2
Started | 119 | 41 | 0
Completed | 119 | 41 | 0
Not Completed | 0 | 0 | 0
Period: Unblinded Phase: From 6 to 12 Months
Arm/Group | BNT162b2 | Placebo | Placebo Then BNT162b2
Started | 119 | 6 (Participants who declined BNT162b2 30 mcg after unblinding.) | 35
Completed | 117 | 3 | 35
Not Completed | 2 | 3 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Other | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention.
Groups:
- BNT162b2: Participants received 2 doses of blinded 30 mcg BNT162b2 vaccine as an intramuscular injection separated by 21 days. Participants were followed up to 12 months after last dose of vaccination.
- Total: Total of all reporting groups
Arm/Group | BNT162b2 | Placebo | Total
Number analyzed (Participants) | 119 | 41 | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.8 (16.16) | 44.8 (17.76) | 46.3 (16.55)
Age, Customized [Count of Participants; unit: Participants]
  20-64 Years | 97 | 33 | 130
  65-85 Years | 22 | 8 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 19 | 79
  Male | 59 | 22 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 119 | 41 | 160
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 119 | 41 | 160
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions by Maximum Severity Within 7 Days After Dose 1
Description: Local reactions included pain at injection site, redness and swelling and were recorded by participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm) and graded as mild: greater than (>) 2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm, severe: >10.0 cm, grade 4 (potentially life threatening): necrosis or exfoliative dermatitis for redness and necrosis for swelling. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity and grade 4 (potentially life threatening): emergency room visit or hospitalization for severe pain. Events were classified as Grade 4 based on study investigator's judgement. Maximum severity was the highest grade within 7 days after vaccination among severity grades where the answers were neither "no" nor missing for at least 1 day.
Time Frame: Within 7 days after Dose 1
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 119 | 41
Percentage of participants
  Redness: Mild | 7.6 [3.5 to 13.9] | 0.0 [0.0 to 8.6]
  Redness: Moderate | 5.9 [2.4 to 11.7] | 0.0 [0.0 to 8.6]
  Redness: Severe | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Redness: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Swelling: Mild | 9.2 [4.7 to 15.9] | 0.0 [0.0 to 8.6]
  Swelling: Moderate | 3.4 [0.9 to 8.4] | 0.0 [0.0 to 8.6]
  Swelling: Severe | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Swelling: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Pain at the injection site: Mild | 57.1 [47.7 to 66.2] | 2.4 [0.1 to 12.9]
  Pain at the injection site: Moderate | 27.7 [19.9 to 36.7] | 0.0 [0.0 to 8.6]
  Pain at the injection site: Severe | 1.7 [0.2 to 5.9] | 0.0 [0.0 to 8.6]
  Pain at the injection site: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]

2. Primary Outcome: Percentage of Participants With Local Reactions by Maximum Severity Within 7 Days After Dose 2
Description: Local reactions included pain at injection site, redness and swelling and were recorded by participants in an e-diary. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm and graded as mild: > 2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm, severe: >10.0 cm, grade 4 (potentially life threatening): necrosis or exfoliative dermatitis for redness and necrosis for swelling. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity, severe: prevented daily activity and grade 4 (potentially life threatening): emergency room visit or hospitalization for severe pain. Events were classified as Grade 4 based on study investigator's judgement. Maximum severity was the highest grade within 7 days after vaccination among severity grades where the answers were neither "no" nor missing for at least 1 day.
Time Frame: Within 7 days after Dose 2
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 116 | 41
Percentage of participants
  Redness: Mild | 6.0 [2.5 to 12.0] | 0.0 [0.0 to 8.6]
  Redness: Moderate | 4.3 [1.4 to 9.8] | 0.0 [0.0 to 8.6]
  Redness: Severe | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Redness: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Swelling: Mild | 4.3 [1.4 to 9.8] | 0.0 [0.0 to 8.6]
  Swelling: Moderate | 4.3 [1.4 to 9.8] | 0.0 [0.0 to 8.6]
  Swelling: Severe | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Swelling: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Pain at the injection site: Mild | 50.9 [41.4 to 60.3] | 0.0 [0.0 to 8.6]
  Pain at the injection site: Moderate | 26.7 [18.9 to 35.7] | 0.0 [0.0 to 8.6]
  Pain at the injection site: Severe | 1.7 [0.2 to 6.1] | 0.0 [0.0 to 8.6]
  Pain at the injection site: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]

3. Primary Outcome: Percentage of Participants With Systemic Events by Maximum Severity Within 7 Days After Dose 1
Description: Systemic events were recorded by participants in e-diary. Fever was categorized as greater than or equal to (>=)37.5 to 38.4 degrees(deg) Celsius(C), >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 hours(h), moderate: >2 times in 24h and severe: required intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h. Events were classified as Grade 4 potentially life threatening (emergency room visit or hospitalization) based on study investigator's judgement. Maximum severity=highest grade within 7 days after vaccination among severity grades where the answers were neither "no" nor missing for at least 1 day.
Time Frame: Within 7 days after Dose 1
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 119 | 41
Percentage of participants
  Fever: >= 37.5 to 38.4 deg C | 11.8 [6.6 to 19.0] | 0.0 [0.0 to 8.6]
  Fever: >38.4 to 38.9 deg C | 2.5 [0.5 to 7.2] | 0.0 [0.0 to 8.6]
  Fever: >38.9 to 40.0 deg C | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Fever: >40.0 deg C | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Fatigue: Mild | 22.7 [15.5 to 31.3] | 7.3 [1.5 to 19.9]
  Fatigue: Moderate | 16.8 [10.6 to 24.8] | 2.4 [0.1 to 12.9]
  Fatigue: Severe | 0.8 [0.0 to 4.6] | 0.0 [0.0 to 8.6]
  Fatigue: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Headache: Mild | 21.8 [14.8 to 30.4] | 7.3 [1.5 to 19.9]
  Headache: Moderate | 10.1 [5.3 to 17.0] | 7.3 [1.5 to 19.9]
  Headache: Severe | 0.8 [0.0 to 4.6] | 0.0 [0.0 to 8.6]
  Headache: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Chills: Mild | 16.0 [9.9 to 23.8] | 4.9 [0.6 to 16.5]
  Chills: Moderate | 8.4 [4.1 to 14.9] | 0.0 [0.0 to 8.6]
  Chills: Severe | 0.8 [0.0 to 4.6] | 0.0 [0.0 to 8.6]
  Chills: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Vomiting: Mild | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Vomiting: Moderate | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Vomiting: Severe | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Vomiting: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Diarrhea: Mild | 3.4 [0.9 to 8.4] | 0.0 [0.0 to 8.6]
  Diarrhea: Moderate | 1.7 [0.2 to 5.9] | 0.0 [0.0 to 8.6]
  Diarrhea: Severe | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Diarrhea: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  New or worsened muscle pain: Mild | 10.1 [5.3 to 17.0] | 2.4 [0.1 to 12.9]
  New or worsened muscle pain: Moderate | 4.2 [1.4 to 9.5] | 0.0 [0.0 to 8.6]
  New or worsened muscle pain: Severe | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  New or worsened muscle pain: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  New or worsened joint pain: Mild | 9.2 [4.7 to 15.9] | 4.9 [0.6 to 16.5]
  New or worsened joint pain: Moderate | 4.2 [1.4 to 9.5] | 0.0 [0.0 to 8.6]
  New or worsened joint pain: Severe | 0.8 [0.0 to 4.6] | 0.0 [0.0 to 8.6]
  New or worsened joint pain: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]

4. Primary Outcome: Percentage of Participants With Systemic Events by Maximum Severity Within 7 Days After Dose 2
Description: Systemic events were recorded by participants in an e-diary. Fever was categorized as >= 37.5 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Fatigue, headache, chills, new or worsened muscle pain and new or worsened joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24h, moderate: >2 times in 24h and severe: required intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h. Events were classified as Grade 4 potentially life threatening (emergency room visit or hospitalization) based on study investigator's judgement. Maximum severity=highest grade within 7 days after vaccination among severity grades where the answers were neither "no" nor missing for at least 1 day.
Time Frame: Within 7 days after Dose 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 116 | 41
Percentage of participants
  Fever: >= 37.5 to 38.4 deg C | 25.0 [17.4 to 33.9] | 0.0 [0.0 to 8.6]
  Fever: >38.4 to 38.9 deg C | 6.9 [3.0 to 13.1] | 0.0 [0.0 to 8.6]
  Fever: >38.9 to 40.0 deg C | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 8.6]
  Fever: >40.0 deg C | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Fatigue: Mild | 25.9 [18.2 to 34.8] | 2.4 [0.1 to 12.9]
  Fatigue: Moderate | 31.0 [22.8 to 40.3] | 0.0 [0.0 to 8.6]
  Fatigue: Severe | 3.4 [0.9 to 8.6] | 0.0 [0.0 to 8.6]
  Fatigue: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Headache: Mild | 25.0 [17.4 to 33.9] | 7.3 [1.5 to 19.9]
  Headache: Moderate | 17.2 [10.9 to 25.4] | 4.9 [0.6 to 16.5]
  Headache: Severe | 1.7 [0.2 to 6.1] | 0.0 [0.0 to 8.6]
  Headache: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Chills: Mild | 24.1 [16.7 to 33.0] | 2.4 [0.1 to 12.9]
  Chills: Moderate | 19.8 [13.0 to 28.3] | 0.0 [0.0 to 8.6]
  Chills: Severe | 1.7 [0.2 to 6.1] | 0.0 [0.0 to 8.6]
  Chills: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Vomiting: Mild | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 8.6]
  Vomiting: Moderate | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Vomiting: Severe | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Vomiting: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Diarrhea: Mild | 5.2 [1.9 to 10.9] | 0.0 [0.0 to 8.6]
  Diarrhea: Moderate | 0.0 [0.0 to 3.1] | 2.4 [0.1 to 12.9]
  Diarrhea: Severe | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  Diarrhea: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  New or worsened muscle pain: Mild | 9.5 [4.8 to 16.3] | 0.0 [0.0 to 8.6]
  New or worsened muscle pain: Moderate | 6.9 [3.0 to 13.1] | 0.0 [0.0 to 8.6]
  New or worsened muscle pain: Severe | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  New or worsened muscle pain: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]
  New or worsened joint pain: Mild | 12.9 [7.4 to 20.4] | 0.0 [0.0 to 8.6]
  New or worsened joint pain: Moderate | 11.2 [6.1 to 18.4] | 0.0 [0.0 to 8.6]
  New or worsened joint pain: Severe | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 8.6]
  New or worsened joint pain: Grade 4 | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 8.6]

5. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Dose 1 up to 1 Month After Dose 2
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Percentage of participants with AEs and the associated 95% confidence interval (CI) based on the Clopper and Pearson method was presented. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were reported in this outcome measure.
Time Frame: Dose 1 up to 1 month after Dose 2
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 119 | 41
Percentage of participants | 10.9 [5.9 to 18.0] | 7.3 [1.5 to 19.9]

6. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) From Dose 1 up to 12 Months After Dose 2
Description: SAE was defined as any untoward medical occurrence that, at any dose, resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect or considered an important medical event. Percentage of participants with SAEs and the associated 95% CI based on the Clopper and Pearson method was presented.
Time Frame: Dose 1 up to 12 months after Dose 2
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 119 | 41
Percentage of participants | 1.7 [0.2 to 5.9] | 0 [0.0 to 8.6]

7. Primary Outcome: Percentage of Participants With Abnormal Hematology and Chemistry Laboratory Values 1 Day After Dose 1 by Age Category
Description: The pre-defined criteria for laboratory parameters included: hemoglobin (HGB), hematocrit, erythrocytes(ery.) less than (<)0.8* lower limit of normal (LLN); ery. mean corpuscular volume, ery. mean corpuscular hemoglobin, ery. mean corpuscular HGB concentration <0.9*LLN and >1.1*upper limit of normal (ULN); platelets <0.5*LLN and >1.75*ULN; leukocytes <0.6*LLN and >1.5*ULN; lymphocytes, neutrophils <0.8*LLN and >1.2*ULN; basophils, eosinophils, monocytes >1.2*ULN; bilirubin >1.5*ULN; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase >3.0*ULN; urea nitrogen, creatinine >1.3*ULN. Percentage of participants with abnormal hematology and chemistry laboratory values by age categories 20 to 64 years and 65 to 85 years were reported in this outcome measure. Categories with at least 1 non-zero data values were reported.
Time Frame: Within 1 day after Dose 1
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention. Here, "Overall Number of Participants Analyzed" signifies participants with at least one result for the laboratory test after study vaccination.
Measure: Number; unit: Percentage of participants
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 9 | 3
Percentage of participants
  20-64 Years: Monocytes | 11.1 | 0.0
  65-85 Years: Lymphocytes | 22.2 | 0.0
  65-85 Years: Monocytes | 11.1 | 0.0
  65-85 Years: Creatinine | 11.1 | 0.0

8. Primary Outcome: Percentage of Participants With Abnormal Hematology and Chemistry Laboratory Values 7 Days After Dose 1 by Age Category
Description: The pre-defined criteria for laboratory parameters included: HGB, hematocrit, ery. <0.8* LLN; ery. mean corpuscular volume, ery. mean corpuscular hemoglobin, ery. mean corpuscular HGB concentration <0.9*LLN and >1.1*ULN; platelets <0.5*LLN and >1.75*ULN; leukocytes <0.6*LLN and >1.5*ULN; lymphocytes, neutrophils <0.8*LLN and >1.2*ULN; basophils, eosinophils, monocytes >1.2*ULN; bilirubin >1.5*ULN; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase >3.0*ULN; urea nitrogen, creatinine >1.3*ULN. Percentage of participants with abnormal hematology and chemistry laboratory values by age categories 20 to 64 years and 65 to 85 years were reported in this outcome measure. Categories with at least 1 non-zero data values were reported.
Time Frame: Within 7 days after Dose 1
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 9 | 3
Percentage of participants
  20-64 Years: Eosinophils | 11.1 | 0.0
  65-85 Years: Lymphocytes | 0.0 | 33.3

9. Primary Outcome: Percentage of Participants With Abnormal Hematology and Chemistry Laboratory Values 7 Days After Dose 2 by Age Category
Description: The pre-defined criteria for laboratory parameters included: HGB, hematocrit, ery. <0.8* LLN; ery. mean corpuscular volume, ery. mean corpuscular hemoglobin, ery. mean corpuscular HGB concentration <0.9*LLN and >1.1*ULN; platelets <0.5*LLN and >1.75*ULN; leukocytes <0.6*LLN and >1.5*ULN; lymphocytes, neutrophils <0.8*LLN and >1.2*ULN; basophils, eosinophils, monocytes >1.2*ULN; bilirubin >1.5*ULN; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase >3.0*ULN; urea nitrogen, creatinine >1.3*ULN. Categories with at least 1 non-zero data value were reported (only 65-85 years: Lymphocytes category was reported).
Time Frame: Within 7 days after Dose 2
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 9 | 3
Percentage of participants | 22.2 | 33.3

10. Primary Outcome: Percentage of Participants With Shift in Hematology and Chemistry Laboratory Values From Baseline to 1 Day After Dose 1 by Age Category
Description: Hematology parameters: hemoglobin, eosinophils, lymphocytes decrease, neutrophil decrease, platelets decrease, white blood cell (WBC) decrease, WBC increase. Chemistry parameters: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, bilirubin increased, creatinine increased, blood urea nitrogen. Laboratory abnormalities were graded by toxicity grading scale for healthy adult volunteers enrolled in preventive vaccine clinical trials as grade 1=mild; grade 2=moderate; grade 3=severe and grade 4=potentially life-threatening. Percentage of participants with shift in hematology and chemistry laboratory values by age categories (20 to 64 years and 65 to 85 years) were reported in this outcome measure. Categories with at least 1 non-zero data values showing any shift in Grade from baseline to 1 day after dose 1 (post-baseline) were reported. Participants whose grade category was unchanged (e.g. normal to normal) were not reported.
Time Frame: From baseline (observation prior to Dose 1) up to 1 day after Dose 1
Population: Safety population included all randomized participants who received at least 1 dose of the study intervention. Here, "Overall Number of Participants Analyzed" signifies participants with at least 1 result for the laboratory test for both baseline and postvaccination visits.
Measure: Number; unit: Percentage of participants
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 9 | 3
Percentage of participants
  20-64 Years- Lymphocytes: Normal (at baseline) to Grade 1 (at post baseline) | 22.2 | 0.0
  20-64 Years- Neutrophil Decrease: Normal (at baseline) to Grade 1 (at post baseline) | 55.6 | 0.0
  20-64 Years- WBC Decrease: Normal (at baseline) to Grade 1 (at post baseline) | 11.1 | 0.0
  65-85 Years- Alanine Aminotransferase Increased: Normal (at baseline) to Grade 1 (at post baseline) | 11.1 | 0.0
  65-85 Years-Aspartate Aminotransferase Increased: Normal (at baseline) to Grade 1 (at post baseline) | 11.1 | 0.0
  65-85 Years- Hemoglobin: Normal (at baseline) to Grade 1 (at post baseline) | 11.1 | 33.3
  65-85 Years- Lymphocytes: Normal (at baseline) to Grade 1 (at post baseline) | 33.3 | 0.0
  65-85 Years- Neutrophil Decrease: Normal (at baseline) to Grade 1 (at post baseline) | 22.2 | 0.0
  65-85 Years- Neutrophil Decrease: Normal (at baseline) to Grade 2 (at post baseline) | 11.1 | 0.0
  65-85 Years- Urea Nitrogen: Normal (at baseline) to Grade 1 (at post baseline) | 0.0 | 33.3
  65-85 Years- WBC Decrease: Normal (at baseline) to Grade 1 (at post baseline) | 33.3 | 0.0

11. Primary Outcome: Percentage of Participants With Shift in Hematology and Chemistry Laboratory Values From Baseline to 7 Days After Dose 1 by Age Category
Description: Hematology parameters included: hemoglobin, eosinophils, lymphocytes decrease, neutrophil decrease, platelets decrease, WBC decrease, WBC increase. Chemistry parameters included: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, bilirubin increased, creatinine increased, urea nitrogen. Laboratory abnormalities were graded by toxicity grading scale for healthy adult volunteers enrolled in preventive vaccine clinical trials as grade 1=mild; grade 2=moderate; grade 3=severe and grade 4=potentially life-threatening. Percentage of participants with shift in hematology and chemistry laboratory values by age categories (20 to 64 years and 65 to 85 years) were reported in this outcome measure. Categories with at least 1 non-zero data values showing any shift in grade from baseline to 7 days after dose 1 (post-baseline) were reported. Participants whose grade category was unchanged (e.g. normal to normal) were not reported.
Time Frame: From baseline (observation prior to Dose 1) up to 7 days after Dose 1
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 9 | 3
Percentage of participants
  20-64 Years- Hemoglobin: Normal (at baseline) to Grade 1 (at post baseline) | 11.1 | 0.0
  20-64 Years- Neutrophil Decrease: Grade 1 (at baseline) to Normal (at post baseline) | 11.1 | 0.0
  65-85 Years- Alanine Aminotransferase Increased: Normal (at baseline) to Grade 1 (at post baseline) | 11.1 | 0.0
  65-85 Years-Aspartate Aminotransferase Increased: Normal (at baseline) to Grade 1 (at post baseline) | 11.1 | 0.0
  65-85 Years- Hemoglobin: Normal (at baseline) to Grade 1 (at post baseline) | 11.1 | 33.3
  65-85 Years- Hemoglobin: Grade 1 (at baseline) to Grade 2 (at post baseline) | 11.1 | 0.0
  65-85 Years- Lymphocytes: Normal (at baseline) to Grade 1 (at post baseline) | 0.0 | 33.3
  65-85 Years- WBC Decrease: Normal (at baseline) to Grade 1 (at post baseline) | 0.0 | 33.3

12. Primary Outcome: Percentage of Participants With Shift in Hematology and Chemistry Laboratory Values From Before Dose 2 to 7 Days After Dose 2 by Age Category
Description: Hematology parameters included: hemoglobin, eosinophils, lymphocytes decrease, neutrophil decrease, platelets decrease, WBC decrease, WBC increase. Chemistry parameters included: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, bilirubin increased, creatinine increased, urea nitrogen. Laboratory abnormalities were graded by toxicity grading scale for healthy adult volunteers enrolled in preventive vaccine clinical trials as grade 1=mild; grade 2=moderate; grade 3= severe and grade 4=potentially life-threatening. Percentage of participants with shift in hematology and chemistry laboratory values by age categories (20 to 64 years and 65 to 85 years) were reported in this outcome measure. Categories with at least 1 non-zero data values showing any shift in grade from before dose 2 to 7 days after dose 2 were reported. Participants whose grade category was unchanged (e.g. normal to normal) were not reported.
Time Frame: Before Dose 2 up to 7 days after Dose 2
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 9 | 3
Percentage of participants
  20-64 Years- Alanine Aminotransferase Increased: Grade 1 (before dose 2) to Normal (post dose 2) | 11.1 | 0.0
  20-64 Years- Eosinophils: Grade 1 (before dose 2) to Normal (post dose 2) | 11.1 | 0.0
  20-64 Years- Hemoglobin: Normal (before dose 2) to Grade 1 (post dose 2) | 11.1 | 0.0
  20-64 Years- Hemoglobin: Grade 1 (before dose 2) to Normal (post dose 2) | 11.1 | 33.3
  20-64 Years- Neutrophil Decrease: Grade 1 (before dose 2) to Normal (post dose 2) | 22.2 | 0.0
  20-64 Years- WBC Decrease: Grade 1 (before dose 2) to Normal (post dose 2) | 11.1 | 0.0
  65-85 Years-Aspartate Aminotransferase Increased: Normal (before dose 2) to Grade 1 (post dose 2) | 11.1 | 0.0
  65-85 Years- Bilirubin: Grade 1 (before dose 2) to Normal (post dose 2) | 11.1 | 0.0
  65-85 Years- Hemoglobin: Normal (before dose 2) to Grade 1 (post dose 2) | 11.1 | 0.0
  65-85 Years- Hemoglobin: Grade 1 (before dose 2) to Grade 2 (post dose 2) | 11.1 | 0.0
  65-85 Years- Lymphocytes: Normal (before dose 2) to Grade 1 (post dose 2) | 0.0 | 33.3
  65-85 Years- Neutrophil Decrease: Normal (before dose 2) to Grade 1 (post dose 2) | 22.2 | 33.3
  65-85 Years- Urea Nitrogen: Normal (before dose 2) to Grade 1 (post dose 2) | 0.0 | 33.3
  65-85 Years- WBC Decrease: Normal (before dose 2) to Grade 1 (post dose 2) | 11.1 | 33.3

13. Primary Outcome: Geometric Mean Titers (GMTs) of SARS-CoV-2 Neutralizing Titers at 1 Month After Dose 2
Description: GMT of SARS-CoV-2 neutralizing titer was calculated by exponentiating the mean logarithm of the titers and the corresponding 95% confidence interval (CI) was based on the Student's t distribution. GMT of SARS-CoV-2 neutralization titer 50% (NT50) was reported in this outcome measure.
Time Frame: 1 month after Dose 2
Population: Evaluable immunogenicity population (EIP): all randomized participants who received 2 doses of the assigned vaccine, with Dose 2 received within the predefined window (within 19-42 days after Dose 1), had at least 1 valid and determinate immunogenicity result from the blood collection within an appropriate window after Dose 2 (within 28-42 days after Dose 2) and had no other major protocol deviations as determined by clinician.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 116 | 41
Titer | 524.5 [459.7 to 598.4] | 10.6 [9.8 to 11.4]

14. Primary Outcome: Geometric Mean Fold Rises (GMFRs) of SARS-CoV-2 Neutralizing Titers From Before Vaccination to 1 Month After Dose 2
Description: GMFR was defined as the result after vaccination divided by the result before vaccination. GMFR and the corresponding 2-sided 95% CIs was calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student's t distribution). GMFR of SARS-CoV-2 NT50 was reported in this outcome measure.
Time Frame: Before vaccination up to 1 month after Dose 2
Population: EIP: all randomized participants who received 2 doses of the assigned vaccine, with Dose 2 received within the predefined window (within 19-42 days after Dose 1), had at least 1 valid and determinate immunogenicity result from the blood collection within an appropriate window after Dose 2 (within 28-42 days after Dose 2) and had no other major protocol deviations as determined by clinician.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 116 | 41
Fold rise | 51.5 [45.2 to 58.7] | 1.1 [1.0 to 1.1]

15. Secondary Outcome: GMTs of SARS-CoV-2 Neutralizing Titers at Baseline, 21 Days After Dose 1; 7 and 14 Days and 6 and 12 Months After Dose 2
Description: GMTs of SARS-CoV-2 neutralizing titers were calculated by exponentiating the mean logarithm of the titers and the corresponding 95% CI was based on the Student's t distribution. GMTs of SARS-CoV-2 NT50 and neutralization titer 90% (NT90) were reported in this outcome measure.
Time Frame: NT50: Baseline (observation prior to Dose 1), 21 days after Dose 1; 7 and 14 days and 6 and 12 months after Dose 2; NT90: Baseline (observation prior to Dose 1), 21 days after Dose 1; 7 and 14 days after Dose 2
Population: EIP: all randomized participants who received 2 doses of the assigned vaccine, with Dose 2 received within the predefined window (within 19-42 days after Dose 1), had at least 1 valid and determinate immunogenicity result from the blood collection within an appropriate window after Dose 2 (within 28-42 days after Dose 2) and had no other major protocol deviations as determined by clinician. "Number Analyzed" signifies participants evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 116 | 41
Titer
  NT50: Baseline | 10.2 [9.8 to 10.6] | 10.0 [10.0 to 10.0]
  NT50: 21 days after Dose 1: number analyzed (Participants) | 116 | 40
  NT50: 21 days after Dose 1 | 29.2 [24.3 to 35.2] | 10.0 [10.0 to 10.0]
  NT50: 7 days after Dose 2 | 408.2 [352.0 to 473.3] | 10.0 [10.0 to 10.0]
  NT50: 14 days after Dose 2 | 379.4 [335.3 to 429.3] | 10.0 [10.0 to 10.0]
  NT50: 6 months after Dose 2: number analyzed (Participants) | 116 | 6
  NT50: 6 months after Dose 2 | 145.6 [126.1 to 168.2] | 20.5 [20.5 to 20.5]
  NT50: 12 months after Dose 2: number analyzed (Participants) | 115 | 3
  NT50: 12 months after Dose 2 | 74.2 [59.6 to 92.3] | 63.8 [0.5 to 8440.7]
  NT90: Baseline | 10.1 [9.9 to 10.2] | 10.0 [10.0 to 10.0]
  NT90: 21 days after Dose 1: number analyzed (Participants) | 116 | 40
  NT90: 21 days after Dose 1 | 11.4 [10.5 to 12.5] | 10.0 [10.0 to 10.0]
  NT90: 7 days after Dose 2 | 104.3 [90.1 to 120.7] | 10.0 [10.0 to 10.0]
  NT90: 14 days after Dose 2 | 95.8 [84.8 to 108.2] | 10.0 [10.0 to 10.0]

16. Secondary Outcome: GMFRs of SARS-CoV-2 Neutralizing Titers Before Vaccination to 21 Days After Dose 1; 7 and 14 Days and 6 and 12 Months After Dose 2
Description: GMFR was defined as the result after vaccination divided by the result before vaccination. GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student's t distribution). GMFRs of SARS-CoV-2 NT50 and NT90 were reported in this outcome measure.
Time Frame: NT50: Before vaccination up to 21 days after Dose 1; 7 and 14 days and 6 and 12 months after Dose 2; NT90: Before vaccination up to 21 days after Dose 1; 7 and 14 days after Dose 2
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 116 | 41
Fold rise
  NT50: before vaccination up to 21 days after Dose 1: number analyzed (Participants) | 116 | 40
  NT50: before vaccination up to 21 days after Dose 1 | 2.9 [2.4 to 3.4] | 1.0 [1.0 to 1.0]
  NT50: before vaccination up to 7 days after Dose 2 | 40.1 [34.6 to 46.5] | 1.0 [1.0 to 1.0]
  NT50: before vaccination up to 14 days after Dose 2 | 37.2 [32.9 to 42.1] | 1.0 [1.0 to 1.0]
  NT50: before vaccination up to 6 months after Dose 2: number analyzed (Participants) | 116 | 6
  NT50: before vaccination up to 6 months after Dose 2 | 14.3 [12.4 to 16.5] | 2.1 [2.1 to 2.1]
  NT50: before vaccination up to 12 months after Dose 2: number analyzed (Participants) | 115 | 3
  NT50: before vaccination up to 12 months after Dose 2 | 7.3 [5.9 to 9.1] | 6.4 [0.0 to 844.1]
  NT90: before vaccination up to 21 days after Dose 1: number analyzed (Participants) | 116 | 40
  NT90: before vaccination up to 21 days after Dose 1 | 1.1 [1.1 to 1.2] | 1.0 [1.0 to 1.0]
  NT90: before vaccination up to 7 days after Dose 2 | 10.3 [8.9 to 12.0] | 1.0 [1.0 to 1.0]
  NT90: before vaccination up to 14 days after Dose 2 | 9.5 [8.4 to 10.7] | 1.0 [1.0 to 1.0]

17. Secondary Outcome: GMTs of SARS-CoV-2 Neutralizing Titers at Baseline, 21 Days After Dose 1; 7 and 14 Days and 1, 6 and 12 Months After Dose 2 in Participants With or Without Confirmed COVID-19 Before Dose 2
Description: GMTs of SARS-CoV-2 neutralizing titers was planned to be calculated by exponentiating the mean logarithm of the titers and the corresponding 95% CI was based on the Student's t distribution.
Time Frame: Baseline (observation prior to Dose 1), 21 days after Dose 1; 7 and 14 days and 1, 6 and 12 months after Dose 2
Population: Data was not analyzed as there were no participants with or without confirmed COVID-19 before Dose 2 prior to unblinding.
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: GMFRs of SARS-CoV-2 Neutralizing Titers Before Vaccination to 21 Days After Dose 1; 7 and 14 Days and 1, 6 and 12 Months After Dose 2 in Participants With or Without Confirmed COVID-19 Before Dose 2
Description: GMFR was defined as the result after vaccination divided by the result before vaccination. GMFRs and the corresponding 2-sided 95% CIs were planned to be calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student's t distribution).
Time Frame: Before vaccination up to 21 days after Dose 1; 7 and 14 days after Dose 2 and 1, 6 and 12 months after Dose 2
Population: as for outcome 17
Arm/Group | BNT162b2 | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Local reactions/systemic events: within 7 days after each dose; SAEs: from Dose 1 up to 12 months after Dose 2 except for Placebo Then BNT162b2 reporting arm; SAEs for Placebo Then BNT162b2 reporting arm: from Dose 3 up to 6 months after Dose 4: other AEs: from Dose 1 up to 1 month after Dose 2 for BNT162b2 and Placebo arms; from Dose 3 up to 1 month after Dose 4 for Placebo Then BNT162b2 reporting arm.
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Systematic events include local reactions and systemic events recorded by participants in e-diary and non-systematic events include all other AEs.
Arm/Group | BNT162b2 | Placebo | Placebo Then BNT162b2
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/41 | 0/35
Serious Adverse Events (participants affected / at risk) | 2/119 | 0/41 | 0/35
Other Adverse Events (participants affected / at risk) | 111/119 | 12/41 | 31/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BNT162b2 (N=119) | Placebo (N=41) | Placebo Then BNT162b2 (N=35)
Pneumonia (Infections and infestations) | 1 | 0 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BNT162b2 (N=119) | Placebo (N=41) | Placebo Then BNT162b2 (N=35)
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 10 | 1 | 0
Chills (CHILLS) (General disorders) | 58 | 3 | 0
Fatigue (FATIGUE) (General disorders) | 75 | 4 | 0
Injection site erythema (REDNESS) (General disorders) | 23 | 0 | 0
Injection site pain (PAIN) (General disorders) | 109 | 1 | 0
Injection site swelling (SWELLING) (General disorders) | 19 | 0 | 0
Pyrexia (FEVER) (General disorders) | 43 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 16
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 35 | 2 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 29 | 1 | 0
Headache (HEADACHE) (Nervous system disorders) | 64 | 8 | 0
Headache (Nervous system disorders) | 2 | 1 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3
Chills (General disorders) | 0 | 0 | 11
Fatigue (General disorders) | 0 | 0 | 21
Injection site erythema (General disorders) | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 31
Injection site pruritus (General disorders) | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 7
Dizziness (Nervous system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs and respective trial sites shall not publish or refer to in writing or orally, in whole or in part, any data, information or materials generated from the study and the services, without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT04588480/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT04588480/SAP_001.pdf